CLINICAL TRIAL: NCT03258879
Title: Comparing the Quality of Labor Analgesia Between Modified Combined Spinal-Epidural and Dural Puncture Epidural Techniques: A Randomized Double Blinded Clinical Trial
Brief Title: Comparison of Labor Analgesia Between Modified Combined Spinal-Epidural and Dural Puncture Epidural Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10017388
Record Dates: First submitted 2017-07-12; First posted 2017-08-23 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: To Determine the Onset of Analgesia (Numerical Rating Scale for Pain = 1) in Minutes
Keywords: Combined spinal epidural analgesia, dural puncture epidural

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified CSE (Experimental): MCSE group: 1 ml of 0.25% bupivacaine will be injected intrathecally
  Interventions: Procedure: Modified CSE
- Dural puncture epidural (Active Comparator): Dural puncture performed with a spinal needle, but no medication will be injected intrathecally.
  Interventions: Procedure: Dural puncture epidural

INTERVENTIONS:
Procedure: Modified CSE — MCSE group: 1 ml of 0.25% bupivacaine will be injected intrathecally
  Arms: Modified CSE
Procedure: Dural puncture epidural — DPE group: Dural puncture performed, but no medication will be injected intrathecally.
  Arms: Dural puncture epidural

SUMMARY:
Epidural, Combined Spinal-Epidural, and more recently dural puncture epidural are forms of neuraxial anesthesia used to provide pain relief in laboring women . The investigators want to assess the onset of pain relief with 2 different neuraxial techniques performed at our center, but which have not yet been compared in the literature: (1) Modified CSE, with only local anesthetic injected into the spinal fluid to reduce side effects of opioids that are seen with the traditional CSE and (2) Dural Puncture Epidural (DPE), involving puncture of the spinal membrane, but without injection of medication into the spinal space. The investigators hypothesize that the onset of labor analgesia will be faster with modified CSE compared to DPE.

DETAILED DESCRIPTION:
Purpose of the research:

* To determine the onset of effective analgesia (Numerical Rating Scale (NRS) for pain </= 1/10 in minutes with the modified CSE and DPE techniques, which is our primary outcome.
* To assess block quality (time to T10 sensory block, motor block, asymmetric block, inadequate block) between the 2 techniques.
* To assess incidence of breakthrough pain as determined by number of physician interventions.
* To determine the incidence of side effects (maternal hypotension, pruritus, nausea, and fetal bradycardia).
* To assess delivery outcomes (vaginal vs. instrumental vs. CS).
* To compare fetal Apgar scores.
* To assess maternal satisfaction with pain relief using Likert scale at 24h.
* To evaluate for potential complications (Post-dural puncture headache, back pain, leg weakness, numbness and infection) related to the techniques at 24h.

Hypothesis:

The investigators hypothesize that the onset of effective analgesia (NRS pain </= 1, in minutes) will be faster with the modified CSE compared to DPE.

Methodology:

Study Design: Randomized Double Blinded Clinical Trial.

Study Implementation:

Once participants are consented for the study, usual care is established with IV cannula insertion, fluid bolus and standard monitors will be applied. Participants will then be randomly assigned into two groups by a computer-generated randomization sequence. Group assignments will be concealed in opaque numbered envelopes and will be opened by the anesthesiologist performing the block immediately before initiation of analgesia. Group 1 will receive a modified combined spinal-epidural (MCSE) and Group 2 will receive a dural puncture epidural (DPE).

The epidural space will be located at the L2-3 or L3-4 interspace using a midline approach with a 17-G, 9 cm Touhy epidural needle using a loss of resistance technique. A single dural puncture with confirmation of free flow of CSF will be performed with a 25-G, 12 cm Whitacre needle placed through the epidural needle. Subsequent intervention varies with the group allocation.

MCSE group: 1 ml of 0.25% bupivacaine will be injected intrathecally DPE group: No medication will be injected intrathecally. Both the groups will subsequently have the epidural catheter placed 4-6 cm into the space and will be checked for a negative aspiration of blood/CSF. In the DPE group, 15 ml of 0.125% bupivacaine will be given as 5ml fractionated boluses. Both groups will have patient controlled epidural analgesia started after the study interventions as follows: Bupivacaine 1.25 mg/mL with fentanyl 2 microgram/ml, background infusion at 8 mL/h, demand dose of 4 mL, lockout interval of 20 minutes.

The anesthesiologist and nurse will be asked not to reveal the group assignment to the patient or study co-investigators so that the patients and the study investigators collecting the data will be blinded to the techniques. The anesthesiologist performing the technique will prepare the medications according to group allocation and will not be involved in any data collection. Attending, fellow or resident anesthesiologists will perform all the techniques.

After block completion, an independent blinded co-investigator will assess the numerical rating scale (NRS) pain scores from 0-10 and other outcomes after the initial dosing, at the 2, 4, 6, 8, 10, 15, 20 and 30 minute marks. The time taken to achieve a NRS equal to or less than 1 will be recorded for all the three groups. Sensory levels will be assessed using ice starting caudad at the S2 dermatome and moving cephalad. Time taken to achieve a block of T10 will be recorded. Patients will be assessed for pruritus and nausea/vomiting every hour, by grading the severity on a scale ranging from 0-3; 0 = none, 1 = mild, 2= moderate and 3 = severe. Motor strength will be assessed hourly with a modified Bromage score (0 = full flexion of knees and ankles, 1 = partial flexion of knees, full flexion of ankles, 2 = inability to flex knees and partial flexion of ankles and 3 = inability to flex knees and ankles). Presence of motor blockade will be defined as modified Bromage score of more than or equal to 1. Following the first 30 minutes, assessments will continue at 60-minute intervals until delivery.

The participant will be monitored for hypotension and fetal bradycardia during this period and up to 1 hour after the procedure. Hypotension is defined as a 20% reduction in the systolic blood pressure from the admission blood pressure in the absence of uterine contraction and will be treated with vasopressors as per the standard of care. Fetal bradycardia is defined as a fetal heart rate of less than 100 beats per minute, persisting for more than 1 minute.

In the event of inadequate analgesia and a unilateral block defined by a difference of more than 2 dermatomal levels between the 2 sides, the participant will be placed on the less blocked side and a supplemental epidural dose will be administered. If the unilateral block persists, the catheter will be withdrawn 1 cm and an additional supplemental epidural dose of 5 ml 2% lidocaine will be given over 2 min. In the event of inadequate analgesia and the presence of inadequate sensory level bilaterally, supplemental epidural dose will be administered. If improvement of analgesia is not observed, the epidural catheter will be replaced.

Mode of delivery and fetal Agar scores will be recorded for all the patients. All the study subjects will be visited on postpartum day 1 and will be assessed for satisfaction with labor analgesia using a Likert scale and any potential complications such as headache, back pain, leg weakness or numbness and paresthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA II healthy adult parturients, at 37-40 weeks gestation with singleton pregnancy and vertex presentation.
* Parturients in early labor with cervical dilatation less than 6 cm requesting epidural analgesia
* Parturients able to provide written informed consent.

Exclusion Criteria:

* Patient refusal to participate in the study.
* Presence of clinically significant disease
* Contraindications to neuraxial analgesia.
* Presence of conditions associated with an increased risk of a cesarean delivery like history of uterine anomaly or surgery, morbid obesity and known fetal anomalies or non-reassuring fetal heart rate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant patients
Enrollment: 80 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of the onset of effective analgesia between the study techniques | 1 year
  Numerical Rating Scale (NRS) for pain </= 1/10 in minutes

SECONDARY OUTCOMES:
Comparison of block quality between the study techniques | 1 year
  Time to T10 sensory block in minutes will be measured
Comparison of the incidence of pruritus between the study techniques | 1 year
  Participants will be assessed for pruritus every hour, by grading the severity on a scale ranging from 0-3; 0 = none, 1 = mild, 2= moderate and 3 = severe
Comparison of the incidence of fetal bradycardia between the study techniques | 1 year
  Fetal bradycardia is defined as a fetal heart rate of less than 100 beats per minute, persisting for more than 1 minute.

CONTACTS AND LOCATIONS:
Overall Officials: Indu Singh, MD, FRCPC, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No